CLINICAL TRIAL: NCT03271983
Title: Evaluation of the Bioavailability of Metronidazole Dermal Products
Brief Title: Pharmacokinetics of Metronidazole Dermal Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00071790
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-03

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- metronidazole gel 1 (Other): RLD gel
  Interventions: Drug: Metronidazole gel 1
- metronidazole gel 2 (Other): generic gel
  Interventions: Drug: Metronidazole gel 2
- metronidazole cream (Other): generic cream
  Interventions: Drug: Metronidazole cream

INTERVENTIONS:
Drug: Metronidazole gel 1 — RLD gel
  Other Names: metronidazole
  Arms: metronidazole gel 1
Drug: Metronidazole gel 2 — generic gel
  Other Names: metronidazole
  Arms: metronidazole gel 2
Drug: Metronidazole cream — generic cream
  Other Names: metronidazole
  Arms: metronidazole cream

SUMMARY:
Generate human PK data by collecting data following the application of metronidazole formulations.

DETAILED DESCRIPTION:
This research study is intended to develop models for in vitro/in vivo correlation (IVIVC) of drug absorption from dermal products. This study will use metronidazole products that have already been approved by the Food and Drug Administration (FDA) and are already sold to customers in the United States; will not include any placebos.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant, women who are of any ethnic background between the age of 18 to 45 years old
2. Subjects must be non-smokers/tobacco users (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches or electronic cigarettes) over the previous 2 months and are not currently using tobacco products
3. Provide written informed consent before initiation of any of the study procedures
4. Agree not to participate in another clinical trial/study during the study period or to participate in an investigational drug study for at least 1 month after the last study session
5. Able to adhere to the study protocol and study restrictions
6. Able to participate in all study sessions
7. Subjects have upper arms large enough to allow for placement of 200 cm2 [31 in2] area for applications of gel or cream. The arm distance from the greater tubercle to the olecranon process should be a minimum of 30 cm. The circumference of the upper arms should be a minimum of 30 cm.
8. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination and medication history
9. Negative urine drug screening test (cannabinoids, amphetamines, barbiturates, benzodiazepine, cocaine, methadone, opiates, PCP)
10. Have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine transaminase (ALT) and aspartate aminotransferase (AST)
11. Have normal screening laboratories for urine protein and urine glucose
12. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of each study session, and must agree to use reliable hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner
13. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 3 months after last study session
14. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute)
15. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-165 mmHg
    * Diastolic blood pressure 60-100 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-20 breaths per minute

Exclusion criteria:

1. Women who are pregnant, lactating, breast feeding or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of the first day of any study session
2. Smokers/tobacco users (current use or use over the previous 2 months of nicotine-containing substances (e.g., cigarettes, cigars, chewing tobacco, gum, snuff, patch or electronic cigarettes)
3. Current participation in any ongoing investigational drug trial/study or clinical drug trial/study
4. History as either reported by the subject or evident to the investigator of infectious disease or skin infection or of chronic skin disease (e.g., psoriasis, atopic dermatitis)
5. History of diabetes
6. History of significant skin cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and did not involve the investigative sites
7. Body Mass Index (BMI) ≥30 kg/m2
8. History of chronic obstructive pulmonary disease or cor pulmonale, or substantially decreased respiratory reserve, hypoxia, hypercapnia or pre-existing respiratory depression
9. Active positive Hepatitis B, C and/or HIV test results
10. Positive urine drug screening test
11. Use of chronic prescription medications during the period 0 to 30 days; or over-the-counter medications (e.g. antihistamines, topical corticosteroids) and short term (<30 days) prescription medications during the period 0-3 days before a study session (vitamins, herbal supplements and birth control medications not included)
12. Currently taking daily anticoagulants (warfarin, heparin, rivaroxaban, dabigatran, etc…) within the past month prior to entry into the study
13. History of blood dyscrasia (abnormal in structure, function and quality)
14. History of Crohn's disease
15. Donation or loss of greater than one pint of blood within 60 days of entry to the study
16. Any prior adverse reaction or hypersensitivity to metronidazole, parabens, other inactive ingredients in the topical gel or cream formulations
17. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study
18. Consumption (food or drink) of alcohol within 48 h prior to dose administration
19. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
20. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application site (upper arms), sunburn, raised moles or scars, open sores at application site (upper arms), scar tissue, tattoo, or coloration that would interfere with placement of metronidazole products, skin assessment, or reactions to metronidazole

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra L Stinchcomb, PhD, Principal Investigator — University of Maryland, Baltimore School of Pharmacy
Locations (1):
- General Clinical Research Center (GCRC) at the University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Metronidazole: Study session 1: metronidazole gel (RLD); followed by at least a one week washout period.
  Study session 2: metronidazole gel (generic); followed by at least a one week washout period.
  Study session 3: metronidazole cream (generic)
Period: Overall Study
Arm/Group | Topical Metronidazole
Started | 7 (The plan was to do n=12 volunteers; however, funding was terminated due to pandemic so only 7 volunteers were completed.)
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Topical Metronidazole
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: PK Parameters
Description: Area under the concentration-time curve from 0 to 25 h
Time Frame: 3 study sessions/subject; each session was 25 h; blood samples obtained at the following time points: -60 min, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 23, 24, 25 h; at least one week washout period between each study session
Measure: Mean (90% Confidence Interval); unit: ng*h/mL
Groups:
- Study Session 1 (RLD Gel): Metronidazole gel: RLD gel
- Study Session 2 (Generic Gel): Metronidazole gel: generic gel
- Study Session 3 (Generic Cream): Metronidazole cream: generic cream
Arm/Group | Study Session 1 (RLD Gel) | Study Session 2 (Generic Gel) | Study Session 3 (Generic Cream)
Number analyzed (Participants) | 7 | 7 | 7
ng*h/mL | 283 [118 to 677] | 341 [226 to 515] | 189 [81.3 to 441]

ADVERSE EVENTS:
Time Frame: For 25 h after product administration plus 72 h after product removal from the arms. Subjects received a phone call within 72 h after completion of the study session to determine there were no adverse events. A total of ~97 h for each study session.
Arm/Group | Study Session 1 (RLD Gel) | Study Session 2 (Generic Gel) | Study Session 3 (Generic Cream)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 2/7 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Session 1 (RLD Gel) (N=7) | Study Session 2 (Generic Gel) (N=7) | Study Session 3 (Generic Cream) (N=7)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
ERYTHEMA (skin reddening) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — from tape used to hold IV in place
Pain at IV site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased blood pressure (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Decreased heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03271983/Prot_SAP_000.pdf